CLINICAL TRIAL: NCT02108769
Title: Induction of Salivary Neuromodulators by Chanting and Breathing Exercise
Brief Title: Yogic Breathing Changes Salivary Components
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Sundaravadivel Balasubramanian, Research Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00024336
Record Dates: First submitted 2014-04-03; First posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Alzheimer Disease; Neurodegenerative Diseases; Cancer
Keywords: Yoga; Yogic breathing; Saliva; Proteomics; Lipdomics; Nerve growth factor; Thirumanthiram
MeSH Terms: conditions — Alzheimer Disease; Neurodegenerative Diseases; Neoplasms; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yogic Breathing (Experimental): 1. Chanting Om
     1. Sharp deep inhalation through nostrils
     2. Slow exhalation through mouth while chanting Om. At this step the subjects will perform a slow and complete exhalation.
     Repeat for 10 min. During the whole period of chanting, the subjects keep their eyes closed.
  2. Yogic Breathing:
     1. Check which of the two nostrils exhibit free flow of air. For the explanation purpose the nostril with free flow of air is treated as Nostril 1 and the other one as Nostril 2.
     2. Close Nostril 2 and inhale a sharp deep breath through Nostril 1 and then close both the nostrils so no inhaled air escapes. Air should not escape through mouth either. This inhalation step should take about 4 seconds.
     3. Hold breath in this position for about 16 seconds.
     4. Open Nostril 2 and exhale for about 8 seconds. Complete exhalation is required. Abdomen will slowly curve-in as the subject exhales. This is normal and encouraged. No air should leak through the Nostril 1 or mouth.
     5. Go to step a).
  Interventions: Behavioral: Yogic Breathing
- Attention Control (Active Comparator): The participants will read a text of their choice for 20 minutes.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Yogic Breathing — 1. Chanting Om
     1. Sharp deep inhalation through nostrils
     2. Slow exhalation through mouth while chanting Om. At this step the subjects will perform a slow and complete exhalation.
     Repeat for 10 min. During the whole period of chanting, the subjects keep their eyes closed.
  2. Yogic Breathing:
     1. Check which of the two nostrils exhibit free flow of air. For the explanation purpose the nostril with free flow of air is treated as Nostril 1 and the other one as Nostril 2.
     2. Close Nostril 2 and inhale a sharp deep breath through Nostril 1 and then close both the nostrils so no inhaled air escapes. Air should not escape through mouth either. This inhalation step should take about 4 seconds.
     3. Hold breath in this position for about 16 seconds.
     4. Open Nostril 2 and exhale for about 8 seconds. Complete exhalation is required. Abdomen will slowly curve-in as the subject exhales. This is normal and encouraged. No air should leak through the Nostril 1 or mouth.
     5. Go to step a).
  Other Names: Pranayama; Moochu Payirchi
  Arms: Yogic Breathing
Behavioral: Attention Control — The participants will read a text of their choice for 20 minutes in a one-on-one session with the Yoga Instructor.
  Other Names: Control
  Arms: Attention Control

SUMMARY:
Our aim is to analyze two ancient Tamil practices (chanting and breathing exercise) if they are capable of stimulating saliva containing agents that can be beneficial to the nervous system. Our study subjects will perform Tamil chanting and Tamil breathing exercise. Saliva will be collected before, during and after the exercises. We will quantify the specific proteins in these salivary samples. The results will benefit further studies in various patient populations.

DETAILED DESCRIPTION:
A. SPECIFIC AIMS

SA1: Obtain a preliminary estimate of the extent to which a structured chanting exercise stimulates salivary secretion that contains quantifiable amounts of NGF in healthy subjects.

SA2: Obtain a preliminary estimate of the extent to which a structured breathing exercise stimulates salivary secretion that contains quantifiable amounts of NGF in healthy subjects.

B. BACKGROUND AND SIGNIFICANCE BACKGROUND Neurodegenerative Diseases Neurodegenerative diseases such as Alzheimer's disease are a major healthcare concern globally. In the USA, AD is the 6th leading cause of death. Both genetic and non-genetic factors contribute to the development of AD. Individuals affected with AD require supports ranging from medications, assisting devices and personal care that pose an enormous emotional and financial burden. AD is associated with significant alterations at the molecular level that eventually translates into cellular, tissue, organ and systemic dysfunction. Therefore, molecular therapy that alters cell functions has been a major clinical option for treating AD . For example, NGF, a trophic factor involved in the development, maintenance and survival of peripheral nervous system and the cholinergic neurons of the central nervous system, show significant reduction in AD subjects. The reduction in NGF causes significant decline in cognitive functions. Therefore administration of NGF is followed as a viable clinical option for AD subjects. In addition to these therapeutic options, non-pharmacological modes of treatment such as meditation and yoga have been considered as alternative approaches to treat AD. Such practices and life-styles are deeply rooted in several ancient cultures. This project is based on two life-style health practices from the ancient Tamil culture.

NGF Nerve growth factor (NGF) is a neurotrophic protein (MW=13 kDa). NGF is produced by every tissue/organ that is innervated by sensory afferents and/or sympathetic efferents, as well as by central (CNS) and peripheral (PNS) nervous system, and immune cells. NGF is important for the functional integrity of cholinergic neurons in CNS and for the development and functional integrity of neurons in PNS. NGF is a survival, differentiation and trophic factor for cells of the immune system and epithelial origin. Salivary glands (submandibular/submaxillary) produce a large amount of NGF in humans and in mice. NGF produced from mouse submaxillary glands is used in several clinical trials. In CNS, NGF is produced in the cortex, the hippocampus and in the pituitary gland; and also in other areas, including the basal ganglia, thalamus, spinal cord and in the retina. NGF binds to its receptor TrkA and activates the mitogenic MAPK, PI3K/Akt and PLC-gamma pathways to mediate cell growth, differentiation and survival. NGF mediated survival is important for the basal forebrain complex (BFC) cholinergic neurons. These neurons contribute to consciousness, memory, attention and arousal. BFC neurons are highly affected in neurodegenerative diseases such as AD. NGF protects BFC neurons in experimental trauma models, and in age-associated cholinergic decline. Due to the positive effects of NGF in multiple systems, development of NGF as a drug is actively pursued for treating neurodegeneration, immune dysregulation, chronic inflammation and autoimmune diseases. However, until recently clinical trials with NGF have been without much success because of hyperalgesia. Recent studies are showing that gene therapy, nasal and ocular routes of NGF administration to be effective with much less nociceptive side effect. Moreover, a recent finding that chemical modification of NGF reduces pain is considered as a new direction in NGF therapy. A Phase II clinical trial assessing the beneficial effects of an adeno-associated virus mediated expression of NGF in the cholinergic neurons of the brain is underway at MUSC involving the co-investigator of this project Dr. Jacobo Mintzer.

NGF is taken up from the target organs by the innervating neurons and transported to axonal body by retrograde axonal transport. Researchers have used quantum-dot labeled NGF to show that each NGF dimer is packaged into individual endosomes during retrograde transport. Retrograde axonal transport of NGF signals for the survival, differentiation, and maintenance of peripheral sympathetic and sensory neurons, and basal forebrain cholinergic neurons. Botulinum toxin follows a retrograde pathway to reach central neurons. Additionally, it was recently confirmed that Botulinum neurotoxins A and E reach distal sites in the nervous system via retrograde long range transport via motor neurons and suggested that this mechanism could be common for the dissemination of other neurotrophic factors as well. This might explain why intranasal application of NGF is considered effective for NGF therapy. In addition, the sublingual route of absorption that bypasses gastrointestinal route is used for the application of nitroglycerine and other psychoactive agents. Thus, our rationale that NGF produced by the salivary glands is taken up by 1) the innervating sensory and motor neurons for retrograde axonal transport to the cell body and transcytosis to reach the central neurons, and 2) the sublingual absorption route into the bloodstream to reach other distal target organs is well within the theoretical framework of production and transport mechanisms established for neuromodulators. It is to be emphasized here that this proposal is the first ever attempt to stimulate NGF by non-invasive methods.

Chanting Chanting and singing are two ancient cultural practices in human history. Recent evidence suggest that these two practices can regulate breathing. The sound symbol Om (Figure 2) is referred as the one-lettered key to happy living. Om is a well-known prefix in several chanting throughout eastern religions. Chanting Om is believed to be associated with physical and emotional well-being. Chanting Om increases the cutaneous peripheral vascular resistance, which is a sign of increased mental alertness even while being physiologically relaxed. In about 40% of Alzheimer's subjects, the middle latency auditory evoked potential (MLAEP) is lacking. Chanting Om is shown to improve MLAEP in normal subjects after chanting suggesting that a similar effect could be observed in AD subjects. Vagal nerve stimulation (VNS) was beneficial in AD subjects as it enhances cognitive functions. Electrical pulsing for VNS showed deactivation of limbic brain regions. Chanting Om also caused a similar deactivation of the limbic brain regions, amygdala, hippocampus, parahippocampal gyrus, insula, orbitofrontal and anterior cingulate cortices and thalamus. The neurophysiological effects of chanting Om could be mediated through the auricular branches of the vagal nerves. However, it is not understood if specific molecular changes, in terms of neurotrophic factors like NGF, occur after Om chanting.

Breathing Exercise Breathing exercise is an active way of regulating breathing. Common breathing frequency is 15 times per minute in normal adult humans. This frequency changes with age and physiological condition. In heart failure subjects Bernardi et al showed that slowing down breathing to be beneficial. Exercises such as yoga, chanting and breathing exercise regulate breathing and cognitive functions. One of the ancient texts referring to the benefits of breathing exercise is Thirumanthiram written by the Tamil sage Thirumoolar whose texts are known for health and longevity practices. Breathing exercise is believed to produce cycles of oxygenation and non-oxygenation states as a means of ischemic preconditioning. Remote ischemic preconditioning, i.e., inducing short periods of ischemia in a remote organ provides protection from a subsequent ischemic insult. Breath-holding increases vagal tone, increases parasympathetic dominance and decreases sympathetic discharges. Regulated breathing leads to predominance in abdominal/diaphragmatic breathing. Thus breathing exercise could be a potential way of inducing ischemic preconditioning in the neurons. It is known in brain and heart that ischemic preconditioning is beneficial in averting future major ischemic events by producing cell survival signaling. Interestingly NGF is a cell survival signaling molecule. Therefore it is conceivable that breathing exercise induces cell survival in central and peripheral nervous system cells via the actions of NGF.

Saliva as a Biomarker A normal human produces about 0.75 to 1.5 L of saliva per day. Saliva contains numerous biologically active molecules including proteins, peptides, mRNA, DNA, and miRNA of both human and oral microbial origin. Salivary secretion regulates the digestive, nervous, immune and respiratory systems. For example, 1) Nerve growth factor (NGF), substance P and calcitonin-gene related peptide (CGRP) are secreted in saliva in response to chronic migraine, and 2) Opiorphin, a potent anti-nociceptive agent is expressed in saliva. Salivary proteomic and mRNA profiling have identified significant differences between control and cancer subjects. These studies indicate that saliva serves as a source of biomarkers in diagnosis and prognosis of a number of pathological conditions including AD.

SIGNIFICANCE Neurodegenerative diseases such as AD constitute a major global healthcare problem. Non-pharmacological and non-invasive practices could alter neurological functions in normal and pathological settings. Salivary secretion of neurotrophic factors indicates that saliva could be a potential source and a biomarker for neurotrophic factors. Therefore, salivary NGF estimation could be a tool for diagnosis and prognosis in AD. Ancient Tamil culture has preserved practices to maintain a healthy psychological and physiological status. Chanting and breathing exercise are known to promote salivary secretion. However, it is not fully understood if such practices induce the expression of neurological factors in the saliva. We aim to quantify salivary NGF in response to chanting and breathing exercise in normal human subjects. This will establish a hitherto unreported relationship between tongue tactile and respiratory signals for salivary secretion of NGF, and its effects on the nervous system. Our project will quantify candidate neurotrophic factor NGF in saliva at basal, during and post-exercise. In future studies we will use proteomic, peptidic and genomic approaches to identify other neurotrophic factors regulated in saliva by these exercises. Our findings will introduce a new paradigm in the treatment and care of individuals with/prone to AD and other neurodegenerative diseases.

Clinical and Translational Impact: Given the fact that AD, aging and other neurodegenerative disorders are associated with declined neurotrophic factor production (e.g. NGF), and that NGF is actively pursued as a drug in clinical trials, our findings that NGF could be stimulated in situ by simple, non-invasive ethnic practices will have strong clinical application. Future studies using genomic and proteomic approaches will identify additional neurotrophic factors in saliva that could potentially be drug targets to treat AD and other neurodegenerative diseases.

C. PRELIMINARY STUDIES None. D. RESEARCH DESIGN AND METHODS Human Subjects

A total of 20 volunteers (male or female), aging 18 and above will be included in the study. The following is a list of conditions for exclusion:

* breathing problems (inability to breath through nostrils, chronic bronchitis, emphysema and asthma)
* speech problems that would prevent chanting
* inability to listen and follow exercise instructions
* sinus congestion
* Sjogren's syndrome
* chronic dry mouth due to medication or other conditions
* use of anti-cholinergic medications Informed consent will be obtained from each subject after completely describing the study.

Human Subject Recruitment Once we get an IRB approval, we will recruit 20 subjects required for this study by posting an advertisement in MUSC elevators and in nearby Yoga centers. Interested participants will contact the PI at the given telephone number. Eligibility of the subjects will be assessed by the PI based on questions given in the Questionnaire. The PI and the participant will agree on an appointment time. The participant will come to the PI's lab at Strom Thurmond Building (STB, Room 222). This meeting room is located on the same floor as the PI's research laboratory. We chose this room for its quiet atmosphere without any interference by other lab personnel during the protocol. This room is reserved via the Gazes Cardiac Research Institute Lab Manager, and is freely available to the PI. Upon arrival, the PI will explain the study to the subject and obtain consent using the Consent Form. The PI will also sign and date the Consent Form and give a copy to the participant. The subject will then fill the Questionnaire to confirm eligibility.

Enrolled and consented subjects will be randomized to one of 2 conditions (the "Chanting/Breathing" (CB) arm versus the "Control" arm. Randomization will be conducted in collaboration with a biostatistician and will be done in a stratified manner (i.e. by gender), to ensure that equal gender distribution in the 2 experimental groups (CB vs. Control). The biostatistician will provide the PI with envelopes containing the study identification number and random group assignment (i.e. CB vs. Control). Each envelope will be opened only after study eligibility has been established and consent has been obtained.

Prior to exercise and sample collection, the PI will teach each subject how to perform chanting and breathing exercise. Each subject will test individually because of ease of sample collection and to avoid any variability that could arise in neuronal stimulation in subjects in the presence of individuals other than the researchers.

Chanting, Breathing exercise and Specimen collection The subjects will get an introduction to the chanting and breathing exercise. As a chanting/yoga/breathing exercise practitioner, the PI will provide this training, which should not take more than 5 minutes to learn. The plan for collecting whole saliva samples is depicted in Figure 3. Salivary samples will be collected once at the beginning of the protocol (Time 0) while the subjects are seated. Saliva will be naturally allowed to accumulate in the oral cavity and the participant will discharge it into the specimen tube (5 mL capacity) with lid.

Chanting Om (C):

The subjects will then chant Om as follows:

1. Sharp deep inhalation through nostrils
2. Slow exhalation through mouth while chanting Om. At this step the subjects will perform a slow and complete exhalation.

These two steps are repeated continuously for 10 min with closed eyes.

Breathing Exercise (BE):

Following the chanting, the subjects will perform the breathing exercise as follows, as instructed by the PI based on Thirumanthiram:

1. Check which of the two nostrils exhibit free flow of air. For the explanation purpose the nostril with free flow of air is treated as Nostril 1 and the other one as Nostril 2.
2. Close Nostril 2 and inhale a sharp deep breath through Nostril 1 and then close both the nostrils so no inhaled air escapes. Air should not escape through mouth either. This inhalation step should take about 4 seconds.
3. Hold breath in this position for about 16 seconds.
4. Open Nostril 2 and exhale for about 8 seconds. Complete exhalation is required. Abdomen will slowly curve-in as the subject exhales. This is normal and encouraged. No air should leak through the Nostril 1 or mouth.
5. Go to step a). During the exercise, if the oral cavity accumulates saliva, the subject can swallow it at the end of exhalation step (Step d). The subjects will perform breathing exercise for 10 min. Salivary samples will be collected at 5 and 10 minutes of breathing exercise in tubes labeled BE-1, BE-2. Thus each individual will provide the following five saliva samples: + (Time 0), Om chanting (C-1 and C2), and Breathing Exercise (BE-1 and BE-2).

Control group In the case of control group, the subjects will sit quietly for the same duration as the CB group. Saliva samples will be collected at the same time points (at 5 min intervals for 20 min) as the CB group.

The approximate total time for the whole protocol will be as follows:

Introduction and Questionnaire - 10 minutes Instruction for chanting, breathing exercise (CB group) or sit quietly (Control group) and salivary sample collection - 10 minutes (CB group) or 5 minutes (Control group) Basal sample collection - 1 minute Om Chanting - 10 minutes Breathing Exercise - 10 minutes Any other question by the subject - 2-3 minutes Total appointment time for a subject = approximately 45 minutes (CB group) 40 minutes (Control group) For the study participants' time and any inconvenience a monetary compensation will be provided.

Processing of samples Place the collected saliva samples on ice. Using sterile techniques, transfer the saliva to centrifuge tubes while measuring the quantity of each sample. The number of samples collected from each sample at each step of the experiment could vary. Treat the samples from individual tubes separately without pooling any sample. Calculate the total volume of saliva during normal resting phase, during chanting and during breathing exercise. Store the samples at -80 degree C until analysis. Samples will be discarded after the data analysis.

Enzyme-linked immunoassay Quantify the levels of NGF in each sample by enzyme-linked immunoassay using commercial kits according to the manufacturer's instructions (Promega). All the reagents necessary to conduct the ELISA experiment are provided in the kit. Additional reagents if any, and the ELISA reader are available to the PI at STB Room 511.

Data management All study data collected from participants by the PI will be entered into a REDCap database, developed with assistance from the project biostatistician. REDCap (Research Electronic Data Capture) is a software toolset and workflow methodology for electronic collection and management of research and clinical trial data available to MUSC researchers. The iterative development and testing process results in a well-planned data collection strategy for individual studies which facilitates data entry, edit checks and eventual statistical analysis. The underlying database is hosted at the MUSC Data Center, and the system is protected behind a login and Secure Sockets Layer (SSL) encryption.

Statistical Analysis Statistical analysis will be done under the guidance of a biostatistician, who has collaborated with the PI in developing this study. Initially, descriptive statistics will be used to characterize the study participants with respect to demographic, any relevant clinical characteristics, and NGF measurements at baseline and over time. Group differences in demographics and other baseline variables will be examined via t-tests, chi square tests, and Fisher's exact tests, as appropriate. This study is meant to obtain preliminary evidence of the effectiveness of these exercises (chanting and/or breathing vs. resting control) to stimulate salivary NGF; as such, no formal hypothesis testing will be conducted. Instead, general linear mixed models (GLMMs) will be used to obtain estimates (and their respective 95% confidence intervals) of the group differences over time with respect to the NGF levels. GLMMs are ideal for analyses involving between- and within-subject variability and are especially useful for repeated measures study designs such as that used for this proposed study. Since age is believed to affect NGF, age will be included as a covariate in all models. Linear, quadratic, and cubic effects of time will be considered. Different types of error covariance structures will be examined, and Akaike Information Criterion values will be used to select the most appropriate-fitting GLMM. Using the GLMM will allow us to characterize the typical trajectory of NGF measurements over time in both experimental conditions and will also afford us the opportunity to compare chanting versus breathing exercises within the CB group. Results from this type of statistical modeling will be valuable for planning (externally funded) future, larger and more definitive studies.

Sample Size Justification Since no formal hypothesis testing will be conducted, statistical power is not relevant for this proposal; thus the sample size justification is based on the precision of our estimation processes and on the learning experiences involved with enrolling, observing, and measuring the subjects in this study as well as conducting the laboratory tests in the most efficient manner as possible. Having n=10 subjects in each experimental group (for a total of n=20 subjects) will allow us to make preliminary estimates of the NGF measurements over time in each group. With n=10 subjects per group, 95% confidence intervals around group mean estimates will extend ~0.6 standard deviations in either direction, and 95% confidence intervals around mean group difference estimates will extend ~0.9 standard deviations in either direction. With n=10 per group, we will also gain a greater understanding of subjects' willingness to be randomized in this type of complementary and alternative medicine study and of the best techniques associated with delivering the chanting and breathing exercises intervention.

E. PROTECTION OF HUMAN SUBJECTS

1. Risks to the Subjects There will be 20 subjects both men and women participating in this study who are in the age group of 18 and above. This protocol will consist of single visit, one-on-one sessions for individual participant. These exercises do not pose any physical, psychological, social risks to the participants. Breach of confidentiality could be one potential risk as the Questionnaire collects health information of the subjects. The participants may feel slightly uncomfortable to spit or drool in the presence of another individual. There is a chance for the participant to feel that they do not know the exercises beforehand or they could feel that they are not fully capable of following the exercise instructions.

   Protections against Risks The instructor will try to make sure that the subjects feel at ease and comfortable. All the information collected in the study will be treated with confidentiality and stored in secured servers as described above. The paper works generated in the present study contains potential personal information.. These documents will be secured in a locked cabinet belonging to the PI located in Room 625 of STB at MUSC. The participants will be identified by an identification number in all the documents, data and in salivary samples. The Informed Consent is the link between the participant identification number and their name. The salivary samples collected will be secured at -80 degree freezer with a lock in STB Room 213 and discarded immediately after the data analysis. The breathing exercises and chanting are mild exercise forms and do not pose any health risks in participants. The study participants will not be contacted for another study.
2. Potential Health Benefits to the Subjects Yogic breathing in particular and yoga in general are good exercises for a healthy life. Several studies indicate that yogic breathing reduces stress and improves the quality of life in multiple patient groups and in otherwise healthy individuals. At the end of the study, the subjects under the Chanting/Breathing Exercise group could feel physically and psychologically better because of the neurotrophic effects. These subjects end up learning new techniques from another culture (cross-cultural experience) to regulate breathing that they can practice daily at their will as continuous practice could benefit them in long run.

ELIGIBILITY:
Inclusion Criteria:

* Anyone

Exclusion Criteria:

* breathing problems (inability to breath through nostrils, chronic bronchitis, emphysema and asthma)
* speech problems that would prevent chanting
* inability to listen and follow exercise instructions
* sinus congestion
* Sjogren's syndrome
* chronic dry mouth due to medication or other conditions
* use of anti-cholinergic medications Informed consent will be obtained from each subject after completely describing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Nerve growth factor quantification | Three months from the date of sample collection
  Nerve growth factor will be quantified by ELISA and Western blotting.

SECONDARY OUTCOMES:
Measuring changes in salivary constituents | 6 months from sample collection
  Western blotting, Multiplex ELISA and Lipidomic analysis will be conducted in saliva samples to determine changes in molecular constituents before and after study exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Sundaravadivel Balasubramanian, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Aloe L, Rocco ML, Bianchi P, Manni L. Nerve growth factor: from the early discoveries to the potential clinical use. J Transl Med. 2012 Nov 29;10:239. doi: 10.1186/1479-5876-10-239. PMID 23190582
- [Background] Kumar S, Nagendra H, Manjunath N, Naveen K, Telles S. Meditation on OM: Relevance from ancient texts and contemporary science. Int J Yoga. 2010 Jan;3(1):2-5. doi: 10.4103/0973-6131.66771. PMID 20948894
- [Background] Rajasekaran R, Narayana A. Thirumular--pioneer of the immunology concept. Bull Indian Inst Hist Med Hyderabad. 2006 Jul-Dec;36(2):129-44. PMID 18175648
- [Derived] Twal WO, Wahlquist AE, Balasubramanian S. Yogic breathing when compared to attention control reduces the levels of pro-inflammatory biomarkers in saliva: a pilot randomized controlled trial. BMC Complement Altern Med. 2016 Aug 18;16:294. doi: 10.1186/s12906-016-1286-7. PMID 27538513
- [Derived] Balasubramanian S, Janech MG, Warren GW. Alterations in Salivary Proteome following Single Twenty-Minute Session of Yogic Breathing. Evid Based Complement Alternat Med. 2015;2015:376029. doi: 10.1155/2015/376029. Epub 2015 Mar 19. PMID 25873979
- See also: South Carolina website for clinical trials. — http://scresearch.org/studies/search?utf8=%E2%9C%93&q=balasubramanian&commit=GO